CLINICAL TRIAL: NCT01797224
Title: Cimzia (Certolizumab Pegol) Pregnancy Exposure Registry: OTIS Autoimmune Diseases in Pregnancy Project
Brief Title: OTIS Cimzia Pregnancy Registry
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: The Organization of Teratology Information Specialists (Other); UCB Pharma (Industry)
Responsible Party: Principal Investigator, Christina Chambers, Professor, Co-Director Center for Promotion of Maternal Health and Infant Development, University of California, San Diego
Other Study IDs: RA0023
Record Dates: First submitted 2012-06-16; First posted 2013-02-22 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Crohn's Disease; Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis; Psoriasis
Keywords: Autoimmune disease; certolizumab pegol; Cimzia; pregnancy; birth defect; birth outcome; TNF; Tumor necrosis factor
MeSH Terms: conditions — Crohn Disease; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Psoriasis; Autoimmune Diseases; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Cohort 1 - Exposed Cohort: Pregnant women with a current diagnosis of an approved indication who have used Cimzia (certolizumab pegol) in the first trimester of pregnancy for any length of time from the date of conception.
- Cohort 2 - Diseased Comparison Cohort: Pregnant women with a current diagnosis of a Cimzia approved indication who have not used Cimzia (certolizumab pegol) during the current pregnancy.
- Cohort 3 - Non-Diseased Comparison Cohort: Pregnant women without a current diagnosis of an autoimmune disease and who have not used Cimzia (certolizumab pegol) at any time in pregnancy, nor have they been exposed to any known human teratogen during pregnancy.
- Group 4 -Cimzia Registry, Not Qualified for the Cohort Study: Women who have used Cimzia (certolizumab pegol) for any length of time following the first day of the last menstrual period until the end of pregnancy who do not qualify for the prospective cohort study.

SUMMARY:
The purpose of the OTIS Autoimmune Diseases in Pregnancy Study is to monitor planned and unplanned pregnancies exposed to certain medications, to evaluate the possible teratogenic effect of these medications and to follow live born infants for five years after birth. With respect to fetal outcome, it is important to evaluate the spectrum of outcomes that may be relevant to a medication exposure during pregnancy, and these include both easily recognizable defects which are visible at birth, as well as more subtle or delayed defects that may not be readily identifiable without special expertise and observation beyond the newborn period.

DETAILED DESCRIPTION:
The purpose of the OTIS Autoimmune Diseases in Pregnancy Project, Cimzia Pregnancy Exposure Registry is to follow pregnant women with or without a Cimzia approved indication who have or have not been treated with Cimzia during pregnancy to evaluate the possible effect of these diseases, and or this medication on the pregnancy outcome including child development and growth up to five years of age.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who reside in the United States or Canada.
Sampling Method: Non-Probability Sample
Enrollment: 925 (Estimated)
Dates: Start 2012-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Major malformations | Duration of pregnancy and up to 1 year of life
  The primary objective of the study is to evaluate the effect of certain medications when used in the first trimester of pregnancy with respect to major structural birth defects.

SECONDARY OUTCOMES:
Minor malformations | At dysmorphological exam which will occur at one time point between birth and 5 years of age
  One secondary objective of the study is to evaluate the effects of certain medications when used in the first trimester of pregnancy with respect to potential minor malformations.
Pregnancy Outcome | Duration of pregnancy and up to 1 year of life
  Another objective of the study is to evaluate the effects of certain medications when used in the first trimester of pregnancy with respect to potential minor malformations
Infant follow-up | Duration of pregnancy and up to 5 years of life
  Pre- and post-natal fetal and infant growth, health and development

CONTACTS AND LOCATIONS:
Overall Officials: Christina Chambers, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- See also: Official Research website of the MotherToBaby/OTIS Studies Coordinated at the University of California, San Diego — https://mothertobaby.org/ongoing-study/cimzia/